CLINICAL TRIAL: NCT01432821
Title: Dopaminergic Reactivity In Idiopathic Generalized Epilepsy: A "Proof Of Concept" Clinical, Pharmacological And Neurophysiological Study
Brief Title: Blinking and Yawning in Epilepsy: The Role of Dopamine
Acronym: BYE BYE DOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C10-27
Record Dates: First submitted 2011-06-14; First posted 2011-09-13 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Generalized Epilepsy
Keywords: Epilepsy,; dopamine; yawning,; blinking eyelids,; electroencephalography
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized; Epilepsy | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apomorphine (Experimental): After randomization healthy volunteers or patients with idiopathic generalized epilepsy receive:
  -sequence A: 1 mg/kg and then 5 mg/kg of apomorphine
  Interventions: Other: Apomorphine (Experimental product)
- Saline (Placebo Comparator): After randomization healthy volunteers or patients with idiopathic generalized epilepsy receive:
  sequence B: 2 injections of saline
  Interventions: Other: Apomorphine (Experimental product)

INTERVENTIONS:
Other: Apomorphine (Experimental product) — Dosage Form: Injection Dosage: 1 or 5 mg / kg
  Route of administration: Subcutaneous
  Duration of treatment: two injections of apomorphine followed by two injections of a placebo one week after or vice versa.
  Two injections will be made by visiting during visits 2 and 3.
  The study was conducted cross-over with two visits EEG recording, the order will be randomized injections:
  * Sequence A during visit 2 followed by sequence B during visit 3
  * or sequence B during visit 2

SUMMARY:
The objective of the present study is to assess dopaminergic reactivity with behavioural markers (i.e. yawning and blinking) in patients with idiopathic generalized epilepsy compared to matched healthy controls, after injection of either low dose of apomorphine or placebo.

Other parameters will be recorded: biochemical (prolactin, GH) and neurophysiological (Spike-Waves Discharge: SWD rating). Safety parameters will be recorded to assess tolerance.

DETAILED DESCRIPTION:
Clinical data regarding the effects of dopaminergic drugs in idiopathic generalized epilepsies are scarce. The general observation that antipsychotic agents (dopaminergic antagonists) worsen seizures, has suggested that dopaminergic agonists would have antiepileptic effects. However, this has never been clearly demonstrated, besides in few limited studies (Mervaala, 1990 ; Quesney, 1980, 1981). More recently, Positron Emission Tomography (PET) investigations using dopaminergic markers (Fluoro-Dopa, SCH23390, DAT) have shown dopaminergic deficits in several epileptic syndromes: ring chromosome 20 syndrome (Biraben 2004), juvenile myoclonic epilepsy (Ciumas 2008), temporal lobe epilepsy (Bouilleret 2008), frontal lobe epilepsy (Fedi 2008). These data give rise to a renewal of interest for the involvement of the dopaminergic neurotransmission in epilepsies. Based on our experimental data from animal studies (see Deransart and Depaulis, 2002), the investigators propose an original study investigating the involvement of the dopaminergic system in idiopathic generalized epilepsies using behavioural as well as neurophysiological markers of the dopaminergic response, in conditions where seizing activities in patients are facilitated (EEG follow-up after sleep deprivation). This approach is based on the concept developed in our laboratory concerning the involvement of the basal ganglia, and more precisely the dopaminergic pathways, in the control of spike-wave discharges in idiopathic generalized epilepsies.

The primary objective is to assess dopaminergic reactivity using a behavioural marker (i.e. yawning) in patients with idiopathic generalized epilepsy compared to matched healthy controls after injection of either low dose of apomorphine or placebo. Other parameters will be recorded as secondary outcomes: behavioural (blinking), biochemical (prolactin, GH) and neurophysiological (Spike-Waves Discharge: SWD rating) markers. Safety parameters will be recorded to assess tolerance.

Experimental data: hyperdopaminergic response in a model of absence-epilepsy in the rat. Since the late 80's, our laboratory has demonstrated the existence of an endogenous neural mechanism that controls the occurrence of epileptic seizures in different animal models, a system based on the hypothesis that the basal ganglia modulate the synchronisation of epileptic rhythmic activities (Depaulis 1994). The studies performed in GAERS (Genetic Absence Epilepsy Rats from Strasbourg, a validated model of absence-epilepsy in rat) have shown that inhibition of the main output structure of basal ganglia (i.e., the substantia nigra pars reticulata) had antiepileptic effects (Depaulis 1994; Deransart 1996). Similarly, deep brain stimulation of the substantia nigra pars reticulata as well as of the subthalamic nucleus interrupts seizures (Vercueil 1998; Feddersen 2007). Systemic and intrastriatal dopamimetics injections in GAERS also suppress seizures, whereas antagonists worsen them (Warter et al, 1988; Deransart et al., 2000). Electrophysiological data showed respectively decreased and increased activity of DA neurons during and at the end of absence-seizures (Lücking et al. 2002). An increase in D3 receptor transcripts was also observed in adult GAERS as compared to inbred non epileptic control rats (NEC), within the ventral striatum (Deransart et al. 2001). These data suggest changes in the DA tone in GAERS with fully developed epileptic phenotype. According to the key role of DA D3 neurotransmission in the foetal cortical development (Levant B, 1995) and modulation of DA tone (Nissbrandt et al., 1995; Gilbert et al., 1995; Kreiss et al., 1995), the researchers investigated whether the putative impaired DA tone in GAERS correlates with functional changes in spontaneous and quinpirole-induced yawning behaviour (Kurashima et al. 1995; Collins et al.2005). The hypothesis of an increased dopaminergic tone in GAERS was thus addressed using pharmacology and microdialysis. In GAERS and NEC (i) spontaneous and quinpirole-induced yawning behaviour and (ii) changes in intra-accumbens dopamine contents induced by amphetamine and K+ and measured by microdialysis were investigated. Spontaneous yawning was significantly decreased in GAERS (0.3±0.2 yawn/hr, n=9) as compared to NEC (5.4±1.2, n=8) and Wistar Harlan rats (9.7±2.3, n=7). Quinpirole-induced yawning was significantly increased in GAERS (29.4±4.9) as compared to NEC (10.5±2.7) and Wistar-Harlan rats (22.6±3.5). Quinpirole also increased the number of absence-seizures in GAERS (+47.4±8.6%). When compared to NEC, basal levels of DA were 40% lower in GAERS whereas amphetamine and K+ produced a higher increase in extracellular dopamine in GAERS. The increased quinpirole-induced yawning in GAERS may account for an overexpression in D3 transcripts. The increased responsiveness of dopamine transmission observed in GAERS after pharmacological manipulations, as compared to NEC, suggests a " hyperdopaminergic " phenotype of GAERS. Altogether, these data support that GAERS have an impaired DA tone that may be associated with the development of mechanisms controlling absences seizures (Deransart et al, in preparation).

Altogether, these data suggest that a phasic involvement (" on request ") of the basal ganglia - notably under the influence of the dopaminergic neurotransmission - may underlie the rapid changes in extracellular activity recorded in output structures of the basal ganglia at the end of seizures in this model (Deransart 2003). Such a phasic functioning of the dopaminergic system in the control of seizures could also reconcile with the apparent discrepancy regarding the fact that seizures appear to escape chronic high-frequency stimulations of the substantia nigra (Feddersen 2007). These data strengthen the need for a re-appraisal of clinical approaches, especially based from a dynamic point of view regarding the involvement of the dopaminergic system in epilepsy.

Clinical data:

* Involvement of the dopaminergic system in idiopathic generalized epilepsies. Exposure to dopaminergic antagonists, like antipsychotic drugs, increases the risk for the patients to display epileptic seizures. The mechanism by which these treatments may lead to such an aggravation remains unknown and, up to date, there is no pharmacological strategy to decrease such a risk. Recent data suggested the involvement of the dopaminergic pathways in several epileptic syndromes: a significant homogeneous decrease in striatal dopamine uptake has been shown using PET in patients with epileptic seizures associated with ring chromosome 20 mosaicism (Biraben, 2004). In this epileptic syndrome, patients display prolonged seizures, reminiscent of an absence status epilepticus. A similar study, using a marker for the dopamine transporter, recently reported a decrease in dopamine re-uptake at the level of the substantia nigra in patients with idiopathic generalized epilepsies (Ciumas, 2008). These data differ from what is observed in neurodegenerative pathologies involving the dopaminergic system (e.g., Parkinson disease) where imaging studies of the dopaminergic transmission show a decrease in synaptic terminals linked to a progressive degenerative process. Data from epileptic patients rather suggest a modulation of the expression of some dopaminergic receptors as well as dynamic changes in the synaptic transmission. In line with our experimental data and the recently published neuroimaging studies, the investigators propose that the reactivity of the dopaminergic system displays special features specific to epileptic patients and may constitute a risk-level marker for epileptic seizures. The conceptual framework of the proposed translationnal study lies on the dynamic involvement of the dopaminergic system and the assessment of its reactivity in epileptic patients.
* Reactivity of the dopaminergic system in idiopathic generalized epilepsies. Low doses of apomorphine, a dopaminergic agonist, induce yawning and palpebral winking in healthy subjects (Blin, 1990). Similarly, higher therapeutic doses induce yawning immediately before therapeutic effect in patients with Parkinson's disease. These data suggest that higher affinity of apomorphine to presynaptic receptor could be involved in promoting yawning and blinking. The study of dopaminergic system response to low doses of apomorphine, below the side-effects threshold (nausea, vomiting, hypotension) represent an original, well-tolerated approach in both patients with epilepsy and healthy subjects. Similar studies have already been published in patients with migraine (Cerbo, 1997) and cocaine users (Colzato, 2008) in order to study dopaminergic reactivity in selected populations. The investigators propose to study dopaminergic reactivity in patients with idiopathic generalized epilepsy compared to matched healthy volunteers, during prolonged EEG after sleep-deprivation, using apomorphine doses of 1 µg/kg and 5 µg/kg. Indeed, apomorphine 0.5 to 2 µg/kg increased spontaneous blinking rate and yawning in healthy volunteers (Blin, 1990). However, a 10 µg/kg dose induced symptoms such as nausea, vomiting, sweating and dizziness in migraineurs (Cerbo, 1997). The study will focus on behaviour (spontaneous and apomorphine-induced yawning and blinking) and EEG (spontaneous and apomorphine induced SWD) as compared to placebo. Prolactin and GH dosing after apomorphine injection will provide a biochemical validation of dopaminergic stimulating effect. Indeed, prolactin secretion is inhibited by dopamine from the hypothalamus, while Growth hormone (GH) is stimulated. Thus, a decrease in prolactin and an increase in GH reflect central dopamine availability. Dosing prolactin and GH response to apomorphine subcutaneous injection represents a way to document the synaptic effects of the drug, as previously described (Aymard, 2003; Friess, 2001).

This project arises from concepts developed in our laboratory from experimental data obtained in an animal model of epilepsy and from recent clinical data from the literature. It aims at improving understanding of dopaminergic transmission dynamics in patients with epilepsy. It could therefore promote the emergence of new markers of susceptibility to epileptic seizures and constitute an opportunity to develop new pharmacological approaches based on dopaminergic neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Men and women aged between 18 and 40
* Person affiliated to social security or beneficiary of such a regime
* idiopathic generalized epilepsy treated with lamotrigine, an association of lamotrigine, topiramate, levetiracetam, lamotrigine or levetiracetam alone (group patients) for at least 14 days without changing doses The idiopathic generalized epilepsy is defined by generalized seizures: generalized tonic-clonic seizures, absences or myoclonic seizures, excluding any other type of seizure, and electroencephalographic appearance following: presence of interictal EEG discharge generalized to type of spikes, spike-wave or wave polyspikes generalized, sporadic or rhythmic> or = 3 Hz background activity is normal.

For healthy volunteers:

* Men and women aged between 18 and 40
* Person affiliated to social security or beneficiary of such a regime

Exclusion Criteria:

* Topic wrongly included
* Deflecting protocol that can skew the primary endpoint
* Primary endpoint missing
* If the investigator considers the health of the subject is incompatible with the continuation of the study.

Criteria for non-inclusion

* For patients:

  * The presence of interictal focal discharges on EEG previous
  * The emergence of partial seizures
  * Restless Leg Syndrome
  * All non-antiepileptic treatment may affect levels of dopamine
  * Current use of illicit drugs.
  * A person deprived of liberty by judicial or administrative person being a measure of legal protection.
  * Pregnant, parturient, lactating mother.
  * For women, lack of effective contraception
* For healthy volunteers:

  * Any medical treatment associated
  * Current use of illicit drugs
  * Pregnant, parturient, lactating mother
  * For women, lack of effective contraception
  * A person deprived of liberty by judicial or administrative person being a measure of legal protection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of yawn | 60 minutes after injections
  Number of yawn at 60 minuts after the injection of apomorphine in patients with idiopathic generalized epilepsy compared to healthy volunteers.
Number of eyelid blinking | 60 minutes after injections
  Number of eyelid Blinking at 60 minuts after the injection of apomorphine in patients with idiopathic generalized epilepsy compared to healthy volunteers.

SECONDARY OUTCOMES:
Number of yawn | at 60 minutes after injections
  Evolution of yawn number between base line period and the 60 minuts following the injection of apomorphine in patients with idiopathic generalized epilepsy compared to healthy volunteers matched.
Number of eyelid blinking in both groups after apomorphin or placebo injection | at 60 minutes after injections
  The number of eyelid blinking after apomorphin or placebo injection is compare in both groups
Neurophysiological assessment of the dopaminergic reactivity | 60 min
  Number and cumulated duration of Spike-waves discharge assessed after injection of apomorphine in patients with idiopathic generalized epilepsy
To test the correlation between the behavioral and neurophysiological markers of dopaminergic reactivity in patients with epilepsy | 60 min
  Correlation between yawning/blinking and the number of Spike-wave discharges in patients with epilepsy (Pearson test)
To assess dopaminergic reactivity with biological markers | 60 min
  Comparison between plasma concentrations of prolactin and growth hormone (GH) in patients and controls after injection of apomorphine or placebo.
Number of Adverse Events as a Measure of Safety and Tolerability | 4 weeks
  This is a descriptive outcome. The number of each adverse event occured at 4 weeks will be listed
Check the absence of spike-wave discharges in healthy volunteers | 60 min
  EEG analysis

CONTACTS AND LOCATIONS:
Overall Officials: Laurent VERCUEIL, Doctor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CIC Department - University Hospital of Grenoble, La Tronche, Isere, France

REFERENCES:
- [Result] Ahmad S, Fowler LJ, Whitton PS. Effect of acute and chronic lamotrigine on basal and stimulated extracellular 5-hydroxytryptamine and dopamine in the hippocampus of the freely moving rat. Br J Pharmacol. 2004 May;142(1):136-42. doi: 10.1038/sj.bjp.0705737. Epub 2004 Mar 22. PMID 15037514
- [Result] Ahmad S, Fowler LJ, Whitton PS. Lamotrigine, carbamazepine and phenytoin differentially alter extracellular levels of 5-hydroxytryptamine, dopamine and amino acids. Epilepsy Res. 2005 Feb;63(2-3):141-9. doi: 10.1016/j.eplepsyres.2005.02.002. PMID 15777732
- [Result] Aymard G, Berlin I, de Brettes B, Diquet B. Pharmacokinetic-pharmacodynamic study of apomorphine's effect on growth hormone secretion in healthy subjects. Fundam Clin Pharmacol. 2003 Aug;17(4):473-81. doi: 10.1046/j.1472-8206.2003.00152.x. PMID 12914551
- [Result] Biraben A, Semah F, Ribeiro MJ, Douaud G, Remy P, Depaulis A. PET evidence for a role of the basal ganglia in patients with ring chromosome 20 epilepsy. Neurology. 2004 Jul 13;63(1):73-7. doi: 10.1212/01.wnl.0000132840.40838.13. PMID 15249613
- [Result] Blin O, Masson G, Azulay JP, Fondarai J, Serratrice G. Apomorphine-induced blinking and yawning in healthy volunteers. Br J Clin Pharmacol. 1990 Nov;30(5):769-73. doi: 10.1111/j.1365-2125.1990.tb03848.x. PMID 2271377